CLINICAL TRIAL: NCT02376231
Title: A Pilot Single Blinded Randomized Controlled Trial to Evaluate the Utility and Efficacy of Neutral Argon Plasma as a New Technology in Achieving Complete Cytoreduction of Advanced Epithelial Ovarian Carcinoma- Initial Feasibility Study
Brief Title: To Evaluate Plasmajet in Achieving Complete Cytoreduction of Advanced EOC- Initial Feasibility Study
Acronym: PJEOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Thumuluru Kavitha Madhuri (Other)
Responsible Party: Sponsor-Investigator, Dr Thumuluru Kavitha Madhuri, Clinical Research Fellow, Royal Surrey County Hospital NHS Foundation Trust
Organization: Royal Surrey County Hospital NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJEOCRSCH
Record Dates: First submitted 2014-05-31; First posted 2015-03-03 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Epithelial Ovarian Cancer
Keywords: EOC Epithelial ovarian cancer; Surgery; nil macroscopic residual disease; Stage 3/4 Epithelial Ovarian Cancer requiring surgery
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Surgical Procedures, Operative; Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Surgery without trial (PJ) device (No Intervention): Standard debulking surgery for EOC without interventional device
- Surgery with trial (PJ) device (Active Comparator): Debulking surgery for EOC with interventional trial device (PJ)
  Interventions: Device: Surgery for EOC with trial (PJ) device (PlasmaJet)

INTERVENTIONS:
Device: Surgery for EOC with trial (PJ) device (PlasmaJet) — Debulking surgery for EOC using PJ device
  Other Names: PlasmaJet device
  Arms: Surgery with trial (PJ) device

SUMMARY:
Surgery for ovarian cancer involves a big cut on your tummy (abdomen) followed by removal of pelvic organs (womb, tubes and ovaries), abdominal organs (fat tissue {omentum}, appendix) and any other tissues involved with cancer. Several studies worldwide have reported that women survive longer and enjoy a longer disease free interval before their disease returns if all visible disease is removed at the time of their surgery. Achieving this is not easy and often there is widespread disease and the surgeons are unable to remove every tumour nodule present as it is attached to the surface of the bowel, diaphragm and other important Extensive surgery with prolonged operating is associated with higher risks. Plasma energy is commonly referred to as the 4th state of matter after solid, liquid and gas. When a gas is heated, it partially or wholly ionizes resulting in high energy particles like ions, electrons and atoms referred to as 'plasma'. PlasmaJet® (PJ) is a new device which uses fine jet of neutral argon plasma from the handpiece that has been shown to have the ability to vaporise nodules close to sensitive organs like the bowel. It may offer the potential to treat the tumour nodules close to sensitive areas like the bowel. There have been no studies exploring its role in vaporising tumour nodules and its impact on survival. The PJ may be used by the surgeon to seal bleeding tissues (coagulate) or to burn away thin layers of tissue (ablate) by vaporization. It is licensed for use to achieve effects of coagulation and ablation. It is similar to conventional surgical devices that are routinely used (called diathermy) to achieve these effects. The PJ however is slightly different in that it may also be used on tissue to vaporise tumour nodules in women with ovarian cancer during surgery though the full extent of this role remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Imaging+/- Clinical +/- laparoscopic e/o pelvic mass and metastatic disease (FIGO III/IV disease) at presentation.
* Confirmation of malignancy on histological/cytological criteria.
* All women aged 18 or over with newly diagnosed FIGO stage III to Stage IV EOC undergoing surgical treatment.
* All women fit to undergo treatment.
* No synchronous malignancy likely to interfere with comparisons.
* Written and informed patient consent

Exclusion Criteria:

* Patient choice
* Patient unfit for any treatment modality
* Patients who are medically unfit for surgery and would only be suitable for chemotherapy.

WITHDRAWAL CRITERIA

* Unforeseen complications in the individual patient will be recorded and then analysed.
* Life threatening situation to the patient, due to any other unrelated complication.
* Patients are free to withdraw from the study at any time with no impact on their care whatsoever.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Ability to achieve complete cytoreduction (nil macroscopic residual disease) either with current standard surgery or using PJ. | At surgery

SECONDARY OUTCOMES:
Per-operative morbidity | 30 days
Post-operative morbidity | 30 days
Bowel resection rate | 6months
Stoma formation rate | 6 months
Disease Free Survival | 3years
Overall Survival | 5 years
Quality of Life | 3 years
  Quality of life based on validated EORTC questionnaires
Cost-effectiveness | 3years
  Measured as an incremental cost per Quality of Life Year (QALY)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynaecological Oncology, Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey, United Kingdom